CLINICAL TRIAL: NCT05217407
Title: A Prospective Clinical Registry Study of Genetic Profiling and Targeted Therapies in Patients With Rare Cancers in ASIA
Brief Title: Marker Assisted Selective ThErapy in Rare Cancers: Knowledge Database Establishing registrY Asia
Acronym: MASTERKEY ASIA
Status: Recruiting | Type: Observational
Sponsor: National Cancer Center, Japan (Other Government)
Responsible Party: Sponsor
Other Study IDs: NCCH2007; 20lk0201002j0001 (Other Grant/Funding Number: AMED)
Record Dates: First submitted 2021-10-24; First posted 2022-02-01 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Rare Malignant Neoplasm
Keywords: Rare cancer; Rare subtype; Registry; Asia; Next-generation sequencing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — whole blood, tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rare cancer: Malignancies with an annual incidence of less than 6 cases per 100,000 population; malignancies categorized as rare cancers in the European RARECARE report; malignancies that are difficult to develop treatments; common cancers with rare tissue subtypes; common cancers that can be regarded as rare based on biological demographics such as age or sex; and cancers of unknow primary are eligible for this study.
  Interventions: Other: Genomic sequence
- Cholangiocarcinoma cohort: This study is a part of MASTER KEY Asia study and designed to be conducted on the patients of cholangiocarcinoma only. The primary endpoint is assigned to the frequency of FGFR2 fusion gene positive cholangiocarcinoma detected by fluorescence in situ hybridization (FISH) in Asian countries. The genetic analysis is performed not only by FISH, but also by next generation sequencing (NGS), so that genetic alterations other than the FGFR2 fusion gene in alterations can be confirmed. To improve outcomes, collecting clinical information is very important to study the relationship between genetic alterations and prognosis, effect of treatments, and the incidence of genomic alterations in cholangiocarcinoma to discover more specific and effective treatment.
  Interventions: Other: Genomic sequence

INTERVENTIONS:
Other: Genomic sequence — Genomic sequence

SUMMARY:
This is a registry study that aims to collect patients' data with advanced-stage rare cancer in Asia-Pacific region. Data includes clinical information, details of treatment, prognosis, pathological diagnosis and genetic biomarkers by next-generation sequencing.

The relationship between cancer types and prognosis, the effect of treatments, and the cancer type-specific incidence of genomic alterations will be investigated to discover more specific and effective treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a histological diagnosis of rare cancer, cancer of unknown primary origin, or cancer of rare tissue subtypes of common cancers. (Defined in protocol.)
2. Patients with Advanced stage cancer.

Exclusion Criteria:

1. Patients with complications of cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Malignancies with an annual incidence of less than 6 cases per 100,000 population; malignancies categorized as rare cancers in the European RARECARE report; malignancies that are difficult to develop treatments; common cancers with rare tissue subtypes; common cancers that can be regarded as rare based on biological demographics such as age or sex; and cancers of unknow primary are eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall incidence of any genomic alteration in overall population | 1 year
  Overall incidence of any genomic alteration in overall population
Overall incidence of any genomic alteration in patients with a certain cancer type | 1 year
  Overall incidence of any genomic alteration in patients with a certain cancer type

SECONDARY OUTCOMES:
Incidence of individual genomic alteration in overall population | 1 year
  The incidence of individual genomic alterations in overall population
Incidence of individual genomic alteration in patients with a certain cancer type | 1 year
  The incidence of individual genomic alterations in patients with a certain cancer type

OTHER OUTCOMES:
Biomarker positive proportion in overall population | 1 year
  The proportion of patients positive for certain biomarkers in overall population
Biomarker positive proportion in patients with a certain cancer type | 1 year
  The proportion of patients positive for certain biomarkers in patients with a certain cancer type
Number of somatic variants within exons in overall population | 1 year
  The number of somatic variants and proportion of variants in overall population
Number of somatic variants within exons in patients with a certain cancer type | 1 year
  The number of somatic variants and proportion of variants in patients with a certain cancer type
Response rate in patients treated with biomarker/genomic alteration-based therapy | 1 year
  Response rate in patients treated with biomarker/genomic alteration-based therapy in overall population, in patients with a certain cancer type, in patients who tested positive/negative for a certain biomarker (any cancer type), in patients with/without a certain genomic alteration (any cancer type), in patients who tested positive/negative for a certain biomarker for a certain cancer type, & in patients with/without a certain genomic alteration for a certain cancer type.
Response rate in patients treated with a therapy other than biomarker/genomic alteration-based therapy | 1 year
  Response rate in patients treated with a therapy other than biomarker/genomic alteration-based therapy in overall population, in patients with a certain cancer type, in patients who tested positive/negative for a certain biomarker (any cancer type), in patients with/without a certain genomic alteration (any cancer type), in patients who tested positive/negative for a certain biomarker for a certain cancer type, & in patients with/without a certain genomic alteration for a certain cancer type.
Response rate in patients treated with immune checkpoint inhibitors | 1 year
  Response rate in patients treated with immune checkpoint inhibitors in overall population, in patients with a certain cancer type, in patients who tested positive/negative for a certain biomarker (any cancer type), in patients with/without a certain genomic alteration (any cancer type), in patients who tested positive/negative for a certain biomarker for a certain cancer type, & in patients with/without a certain genomic alteration for a certain cancer type.
Disease control rate in patients treated with biomarker/genomic alteration-based therapy | 1 year
  Disease control rate in patients treated with biomarker/genomic alteration-based therapy in overall population, in patients with a certain cancer type, in patients who tested positive/negative for a certain biomarker (any cancer type), in patients with/without a certain genomic alteration (any cancer type), in patients who tested positive/negative for a certain biomarker for a certain cancer type, & in patients with/without a certain genomic alteration for a certain cancer type.
Disease control rate in patients treated with a therapy other than biomarker/genomic alteration-based therapy | 1 year
  Disease control rate in patients treated with a therapy other than biomarker/genomic alteration-based therapy in overall population, in patients with a certain cancer type, in patients who tested positive/negative for a certain biomarker (any cancer type), in patients with/without a certain genomic alteration (any cancer type), in patients who tested positive/negative for a certain biomarker for a certain cancer type, & in patients with/without a certain genomic alteration for a certain cancer type.
Disease control rate in patients treated with immune checkpoint inhibitors | 1 year
  Disease control rate in patients treated with immune checkpoint inhibitors in overall population, in patients with a certain cancer type, in patients who tested positive/negative for a certain biomarker (any cancer type), in patients with/without a certain genomic alteration (any cancer type), in patients who tested positive/negative for a certain biomarker for a certain cancer type, & in patients with/without a certain genomic alteration for a certain cancer type.
Overall survival | 1 year
  Overall survival in overall population, in patients with a certain cancer type, in patients who tested positive/negative for a certain biomarker (any cancer type), in patients with/without a certain genomic alteration (any cancer type), in patients who tested positive/negative for a certain biomarker for a certain cancer type, & in patients with/without a certain genomic alteration for a certain cancer type.
Progression-free survival | 1 year
  Progression-free survival in overall population, in patients with a certain cancer type, in patients who tested positive/negative for a certain biomarker (any cancer type), in patients with/without a certain genomic alteration (any cancer type), in patients who tested positive/negative for a certain biomarker for a certain cancer type, & in patients with/without a certain genomic alteration for a certain cancer type.
Proportion of patients receiving no treatment with observation-only in real-world clinical practice | 1 year
  Proportion of patients receiving no treatment with observation-only in real-world clinical practice in overall population & in patients with a certain cancer type. Proportion of patients receiving no treatment or observation with best supportive care in real-world clinical practice in overall population & in patients with a certain cancer type.

CONTACTS AND LOCATIONS:
Overall Officials: Noboru Yamamoro, MD, PhD, Principal Investigator — National Cancer Center Hospital, Japan; Kan Yonemori, MD, PhD, Study Director — National Cancer Center Hospital, Japan; Kenichi Nakamura, MD, PhD, Study Director — National Cancer Center Hospital, Japan; Yuta Maruki, MD, Study Director — National Cancer Center Hospital, Japan; Takuji Okusaka, MD, PhD, Principal Investigator — National Cancer Center Hospital, Japan
Locations (18):
- National Cancer Center Hospital, Japan, Chuo-ku, Tokyo, Japan
- Malaysia (6):
  - Hospital Sultan Ismail, Johor Bahru, Johor
  - Hospital Pulau Pinang, Pulau Pinang, Pulau Pinang
  - Sarawak General Hospital, Kuching, Sarawak
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Center, Kuala Lumpur
  - Institut Kanser negara, Putrajaya
- St. Luke's Medical Center, Manila, Philippines
- National Cancer Center Korea, Seoul, South Korea
- Taiwan (2):
  - National Taiwan University Hospital, Taipei, Zhongzheng
  - Taipei Veterans General Hospital, Taipei
- Thailand (5):
  - Mahidol University by Faculty of Medicine, Ramathibodi Hospita, Bangkok
  - Mahidol University by Faculty of Medicine, Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Faculty of Medicine, Prince of Songkla University, Hat Yai
  - Khon Kaen University by Faculty of Medicine, Srinagarind Hospital, Khon Kaen
- Vietnam (2):
  - National Cancer Vietnam, Hanoi
  - Ho Chi Minh City Oncology Hospital, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Okuma HS, Yonemori K, Narita SN, Sukigara T, Hirakawa A, Shimizu T, Shibata T, Kawai A, Yamamoto N, Nakamura K, Nishida T, Fujiwara Y. MASTER KEY Project: Powering Clinical Development for Rare Cancers Through a Platform Trial. Clin Pharmacol Ther. 2020 Sep;108(3):596-605. doi: 10.1002/cpt.1817. Epub 2020 Apr 7. PMID 32112563